CLINICAL TRIAL: NCT06390514
Title: The Benefits of Vibrating Floors for Deaf Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PLANCHER
Record Dates: First submitted 2024-01-08; First posted 2024-04-30 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Deaf Children
Keywords: vibrating floor benefits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with the vibrating floor (Experimental)
  Interventions: Other: vibrating floor; Other: No vibrating floor
- without the vibrating floor (Active Comparator)
  Interventions: Other: vibrating floor; Other: No vibrating floor

INTERVENTIONS:
Other: vibrating floor — activities with vibrating floor
Other: No vibrating floor — activities without vibrating floor

SUMMARY:
In view of the difficulties observed in the oral language development of deaf children, it is essential to offer them appropriate and effective care as early as possible. One of the modalities frequently used clinically to stimulate this perception of language in the deaf child is to use the tactile sense via vibrations. One such tactile tool used by speech therapists is the vibrating floor, which enables the child to feel sounds through the vibrations perceived by his or her body. Although used in many institutions, there is very little scientific evidence to date of the effectiveness of using the vibrating floor with deaf children.

ELIGIBILITY:
Inclusion Criteria:

* Deaf children whose project is to develop oral French language skills
* Deaf children with cochlear implants or hearing aids
* Children with previous experience of the vibrating floor

Exclusion Criteria:

* intellectual disability
* impairment

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Language assessment | Throughout the entire study, approximately during 24 months
  sound detection, discrimination and repetition

SECONDARY OUTCOMES:
Questionnaire on feelings and well-being | Throughout the entire study, approximately during 24 months
  feelings about vibrating floor

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bragard, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Bragard Anne, Louvain-la-Neuve, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No